CLINICAL TRIAL: NCT02499432
Title: Improving Implementation of Evidence Based PTSD Psychotherapy for Veterans in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: The Tug McGraw Foundation (Unknown)
Responsible Party: Principal Investigator, Carie Rodgers, Staff Psychologist, Veterans Medical Research Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 12-1061
Record Dates: First submitted 2012-11-29; First posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: PTSD
Keywords: Evidence Based Psychotherapy; Implementation; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Enhancement (Experimental): Motivational Interviewing/Enhancement is a form of collaborative discussion for strengthening motivation and commitment to change.
  Interventions: Behavioral: Motivational Enhancement
- Standard training (No Intervention): Training as usual

INTERVENTIONS:
Behavioral: Motivational Enhancement — Motivational Enhancement/Interviewing is a form of discussion that seeks to increase change behavior.
  Other Names: Motivational Interviewing
  Arms: Motivational Enhancement

SUMMARY:
To further increase the access of evidence based psychotherapies for Veterans with Posttraumatic Stress Disorder, we propose to offer training and intensive consultation to community-based providers in Cognitive Processing Therapy for Posttraumatic Stress Disorder. However, we believe that many clinicians may not implement Cognitive Processing Therapy or take advantage of consultation after initial training. For this reason, we propose to examine the effectiveness of an enhanced training method, which would add Motivational Interviewing to the standard Cognitive Processing Therapy training. Motivational Interviewing is a form of collaborative discussion for strengthening motivation and commitment to change. We hypothesize that augmenting the standard Cognitive Processing Therapy training with these techniques will reduce providers' reluctance to fully implement the interventions.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* currently licensed in their mental health discipline or a graduate level trainee in their mental health discipline

Exclusion Criteria:

* Have completed a 2-day training in Cognitive Processing Therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change assessed by Evidence Based Practice Attitudes Scale - 50 | immediately pre-intervention/immediately post 2 day intervention/6 month followup
  Pre intervention will be evaluated immediately before the 2 day training begins and post intervention will be evaluated immediately following the training. Followup will be collected approximately 6 monte after post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Carie S Rodgers, PhD, Principal Investigator — San Diego VA Healthcare System/UCSD/VMRF
Locations (1):
- Veterans Medical Research Foundation, San Diego, California, United States